CLINICAL TRIAL: NCT04280744
Title: Feasibility of a Music Therapy Intervention to Decrease Stress During Pediatric Critical Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Jessica Jarvis, Postdoctoral Scholar, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY19100263
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Critical Illness; Hypoxia, Brain
MeSH Terms: conditions — Critical Illness; Hypoxia, Brain | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Single-arm feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music therapy (Experimental): Music listening intervention provided by a board certified music therapist.
  Interventions: Other: Music therapy

INTERVENTIONS:
Other: Music therapy — Patient preferred song will be provided in a sedative manor (e.g., 60-80 beats per minute) using live music (singing with guitar accompaniment) by a board certified music therapist.
  Other Names: Music listening

SUMMARY:
Admission into a pediatric intensive care unit (PICU) is a highly stressful experience for child and family. High levels of stress can negatively impact outcomes, yet non-pharmacological interventions to decrease stress in the PICU are severely lacking. This is a prospective, single-arm feasibility trial that will explore the feasibility and acceptability of a music therapy intervention to decrease stress in the PICU among families of children receiving invasive or noninvasive mechanical ventilation.

Objectives: The aims of this study are to: 1) Assess the feasibility of implementing a music therapy intervention in the PICU among children receiving invasive or non-invasive mechanical ventilation; 2) Determine the acceptability of the music therapy intervention in the ICU among caregivers, patients, and pediatric and cardiac ICU staff; 3) Explore the variability in child and caregiver stress outcomes throughout ICU admission. Hypothesis: The music therapy intervention will be feasible, as determined by recruitment, retention, protocol adherence, and data collection rates, and will be acceptable to participants and to PICU staff.

Sample: This study will recruit 20 families that include children aged 2 months - 17 years old admitted with an expected length of ICU stay greater than 72 hours. Of these 20 families, the investigators will specifically recruit 10 families whose child is admitted for a hypoxic brain injury. Eligible children are receiving either noninvasive mechanical ventilation (i.e., continuous or bilevel positive airway pressure), invasive mechanical ventilation, or have an established tracheostomy tube and with escalated support settings. One primary caregiver will be enrolled along with the child admitted into the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Parent/caregiver aged 18 years or older.
* Children aged 2 months - 17 years admitted to the PICU with an expected length of stay greater than 72 hours
* Child is receiving either noninvasive mechanical ventilation (i.e., continuous or bilevel positive airway pressure), invasive mechanical ventilation, or have an established tracheostomy tube and with escalated support setting

Exclusion Criteria:

* The legal guardian is unclear,
* Caregiver does not read, write, and speak English
* Child is not expected to survive that PICU stay or has care limitations in place
* Child has deafness in both ears, in foster care or justice system, or experiences musicogenic epilepsy.

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of participant recruitment | Throughout study completion, anticipated 1 year
  Feasibility of participant recruitment will be determined via recruitment rate
Feasibility of participant retention | Post-intervention completion, anticipated 2 weeks
  Feasibility of participant retention will be determined via retention
Feasibility of protocol | Throughout study completion, anticipated 1 year
  Feasibility of protocol will be determined via percentage of sessions that adhere to protocol
Feasibility of data collection | Throughout study completion, anticipated 1 year
  Feasibility of data collection will be determined via percentage of participants with complete data capture
Acceptability of intervention among participants | Post-intervention, anticipated 2 weeks
  Acceptability will be assessed via interviews with participants (caregivers and children 8 years and older) to ascertain intervention benefits, barriers, and potential optimizations.

SECONDARY OUTCOMES:
Change in heart rate | Throughout intervention completion, anticipated 2 weeks
  Change in child participant heart rate during intervention
Change in oxygen saturation | Throughout intervention completion, anticipated 2 weeks
  Change in child participant oxygen saturation during intervention
Change in blood pressure | Throughout intervention completion, anticipated 2 weeks
  Change in child participant blood pressure during intervention
Change in saliva cortisol | Throughout intervention completion, anticipated 2 weeks
  Change in child and caregiver participant saliva cortisol levels pre-post intervention
Change in saliva inflammatory biomarkers | Throughout intervention completion, anticipated 2 weeks
  Change in child participant saliva inflammatory biomarker levels pre-post intervention
Visual Analog Scale - Anxiety | Throughout intervention completion, anticipated 2 weeks
  Change in caregiver participant self-reported anxiety pre-post intervention. 0-100, higher score indicates greater anxiety level.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Jarvis, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bradt J, Dileo C. Music interventions for mechanically ventilated patients. Cochrane Database Syst Rev. 2014;2014(12):CD006902. doi: 10.1002/14651858.CD006902.pub3. Epub 2014 Dec 9. PMID 25490233
- [Background] Chlan LL, Weinert CR, Heiderscheit A, Tracy MF, Skaar DJ, Guttormson JL, Savik K. Effects of patient-directed music intervention on anxiety and sedative exposure in critically ill patients receiving mechanical ventilatory support: a randomized clinical trial. JAMA. 2013 Jun 12;309(22):2335-44. doi: 10.1001/jama.2013.5670. PMID 23689789
- [Background] Liu MH, Zhu LH, Peng JX, Zhang XP, Xiao ZH, Liu QJ, Qiu J, Latour JM. Effect of Personalized Music Intervention in Mechanically Ventilated Children in the PICU: A Pilot Study. Pediatr Crit Care Med. 2020 Jan;21(1):e8-e14. doi: 10.1097/PCC.0000000000002159. PMID 31652195